CLINICAL TRIAL: NCT04934917
Title: Brain Imaging of Pain-Related Processing and Structural Properties in Disc Degenerative Disease
Acronym: POADOSpre
Status: Terminated | Type: Observational
Why Stopped: Covid related problems
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Kosek, Principal Investigator, Professor, MD, Karolinska Institutet
Other Study IDs: 2019-01142_1pre
Record Dates: First submitted 2021-05-25; First posted 2021-06-22 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with disc degenerative disease (DDD): Patients suffering from disc degenerative disease, age 30-60 years that are on the waiting list for surgery (fusion/disc implants) at Stockholm Spine Center, Stockholm, Sweden.
  Interventions: Device: Magnetic Resonance Imaging
- Healthy controls (HC): Healthy controls matched according to age and sex, no chronic pain conditions.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Magnetic Resonance Imaging. Pain testing: Temporal summation, Pain thresholds. Assessment of symptoms: Questionnaires. All interventions are made at baseline only (1 time/subject).

SUMMARY:
In this study, we apply brain MR imaging techniques at 3 Tesla to assess pain-relevant processing in patients with disc degenerative disease (DDD) scheduled for back surgery and age- and gender-matched controls without back pain. Data collection pre-surgery is performed over two days: On the first day, all participants undergo a battery of questionnaires relevant for individuals with chronic pain and pain sensitivity testing, including temporal summation and pressure pain thresholds. On the second day, participants undergo a MRI protocol, which includes functional MRI (fMRI) and diffusion tensor imaging to assess microstructural properties and structural connectivity. During fMRI, an experimental pressure pain paradigm is performed at the calf i.e. a location not connected to patients' chronic pain condition. Instead, the experimental pain paradigm serves as a condition to test processing of noxious stimulation unrelated to patients' experienced chronic pain. The noxious input pressure is individually calibrated to 50 on a 0-100 VAS scale to ensure that individual pain perceptions, despite different pressure intensities, are comparable across participants. The sensory stimulation will consist of a low standardized pressure intensity (150kPa). In an additional fMRI paradigm, participants do not receive stimulation but are instructed to continuously rate fluctuating spontaneous ongoing back pain (DDD) or perceived unpleasantness (controls).

This project aims at investigating measures of brain architecture, neural response connected with evoked pain, connectivity (structural and functional) and pain-relevant psychometrics and questionnaire data in disc degenerative disease patients scheduled for back surgery. Specifically, MRI is performed to test whether i) patients display differences in properties of the mesolimbic circuit compared to healthy individuals and ii) behavioural as well as clinical characteristics related to the acquired MRI markers. This study is intended to serve as a baseline in a longitudinal project testing associations with between findings at baseline and following surgery (fusion/disc implants).

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria:

* 30-60 year
* Right-handed
* DDD patients: Radiologically verified DDD and DDD pain as their main pain complaint

Exclusion Criteria:

* previous spine surgery
* significant pain problems due to other causes and/or other chronic pain syndromes
* inflammatory rheumatic diseases
* neurological/psychiatric disorders
* severe cardiovascular disease
* substance abuse
* BMI>40
* Contraindication to MRI

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited through clinical collaborators (Stockholm Spine Center, Rygg Kirurgisk Centrum); HC will be recruited via online advertisement on the institution's website
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (rsfMRI) | Baseline
  Analysis of network connectivity during resting state
Functional magnetic resonance imaging (BOLD) | Baseline
  cerebral pain related activation following evoked pressure pain stimuli
Diffuse Tensor Imaging | Baseline
  White matter microstructure (e.g. structural connectivity)
Pressure pain thresholds | Baseline
  Pressure allometry (mmHg)
Temporal summation | Baseline
  Pain ratings during repeated pressure stimuli, ratings from 0-100, with 100 being worst pain imaginable

SECONDARY OUTCOMES:
Pain intensity ratings | Baseline
  Visual analogue scale, 0-100 mm, 100 mm, worst possible pain
Oswestry Disability Index | Baseline
  0-100, 0=no disability, 100= worst disability
Fibromyalgia criteria-2016 revision (American College of Rheumatology) | Baseline
  Calculation of FMness score, 0-31, 0 = no symptoms, 31 = worst symptoms
Multidimensional Fatigue Inventory | Baseline
  Total fatigue score, range 20-100, 100 = worst fatigue
Pain catastrophizing scale | Baseline
  Total score 0-52, high values more catastrophizing
Beck Depression Inventory | Baseline
  Scores 0-63, with 63 highest depression
State-Trait Anxiety Inventory | Baseline
  Scores 20-80 for state and 20-80 for trait anxiety, higher levels indicate more anxiety
EuroQual-5D | Baseline
  Scale ranging from -0.224 to 1, with 1 being highest possible health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kosek, Prof, MD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institute, Stockholm
  - Karolinska Insitutet, Stockholm

IPD SHARING:
Plan to Share IPD: No